CLINICAL TRIAL: NCT05876442
Title: Efficacy of Extracorporeal Shock Wave Therapy Plus High-Intensity LaserTherapy on Carpal Tunnel Syndrome Post Burn Injury.
Brief Title: Efficacy of EPSW Plus HILT on Carpal Tunnel Syndrome Post Burn Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004498
Record Dates: First submitted 2023-05-12; First posted 2023-05-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Burn Injury
Keywords: Extracorporeal shock wave therapy; High Intensity Laser Therapy; Carpal Tunnel Syndrome
MeSH Terms: conditions — Burns; Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: ESWT plus HILT in addition to Traditional Physical Therapy Exercise . (Experimental): patients will receive Extraporeal Shock wave therapy at the area of the wrist for 5 minutes 1 time a week for 2 months, then High-intensity laser therapy at the site of the carpal bones for 5 minutes 2 times a week. Then a program of traditional physical therapy exercises for post-burn carpal tunnel syndrome for 30 minutes of stretching exercise for the wrist and carpal region with the fingers flexed and extended. Followed by strengthening exercises for the wrist flexors, extensors, radial and ulnar deviation muscles. Mobilizing exercise, tendon gliding exercise, and instructed to wear a wrist splint at night.
  Interventions: Device: Extracorporeal Shock Wave Therapy.; Device: High Intensity Laser Therapy; Other: Traditional Physical Therapy Exercise Program
- Experimental: Group B: ESWT plus Traditional Physical Therapy Exercise . (Experimental): Patients will receive Extraporeal Shock wave therapy at the area of the wrist for 5 minutes 1 time a week for 2 months, Then a traditional physical therapy exercise program for the post-burn carpal tunnel syndrome for 30 minutes of stretching exercise for the wrist and carpal region with the fingers flexed and extended. They were followed by strengthening exercises for the wrist flexors, extensors, and radial and ulnar deviation muscles. Mobilizing exercise, tendon gliding exercise, and instructed to wear a wrist splint at night
  Interventions: Device: Extracorporeal Shock Wave Therapy.; Other: Traditional Physical Therapy Exercise Program
- Experimental: Group C:HILTplus Traditional Physical Therapy Exercise. (Experimental): patients will receive High-intensity laser therapy at the area of the carpal bones for 5 minutes 2 times a week for 2 monthes. Then a program of traditional physical therapy exercises for post-burn carpal tunnel syndrome for 30 minutes of stretching exercise for the wrist and carpal region with the fingers flexed and extended. Followed by strengthening exercises for the wrist flexors, extensors, and radial and ulnar deviation muscles. Mobilizing exercise, tendon gliding exercises, and instructed to wear a wrist splint at night
  Interventions: Device: High Intensity Laser Therapy; Other: Traditional Physical Therapy Exercise Program
- Traditional Physical Therapy Exercise. (Active Comparator): patients will receive a program of traditional physical therapy exercise for post-burn carpal tunnel syndrome for 30 minutes of stretching exercise for the wrist and carpal region with the fingers flexed and extended. They were followed by strengthening exercises for the wrist flexors, extensors, and radial and ulnar deviation muscles. Mobilizing exercise, tendon gliding exercise, and instructed to wear a wrist splint at night.
  Interventions: Other: Traditional Physical Therapy Exercise Program

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy. — Patients will receive EPSW therapy at the area of the wrist for 5 minutes 1 time a week for 2 months.
  Arms: Experimental: Group B: ESWT plus Traditional Physical Therapy Exercise .; Group A: ESWT plus HILT in addition to Traditional Physical Therapy Exercise .
Device: High Intensity Laser Therapy — High-intensity laser therapy at the area of the carpal bones for 5 minutes 2 times a week for two months..
  Arms: Experimental: Group C:HILTplus Traditional Physical Therapy Exercise.; Group A: ESWT plus HILT in addition to Traditional Physical Therapy Exercise .
Other: Traditional Physical Therapy Exercise Program — 30 minutes of stretching exercise for the wrist and carpal region with the fingers flexed and extended. Followed by strengthening exercises for the wrist flexors, extensors, and radial and ulnar deviation muscles. Mobilizing exercise, tendon gliding exercise, and instructed to wear a wrist splint at night for two months.

SUMMARY:
To study the effect of adding ESWT as a noninvasive short-term treatment plus high-level laser therapy for moderate carpal-tunnel syndrome post-burn injuries.

DETAILED DESCRIPTION:
To study the effect of adding ESWT as a noninvasive short-term treatment plus high-level laser therapy for mild to moderate carpal tunnel syndrome post-burn injuries.

The effects of combining EPSW with High-intensity Laser Therapy for improving pain, Symptoms and function of motion, muscle strength, and quality of life in inpatients with carpal tunnel syndrome post-burn injuries

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with carpal tunnel syndrome after thermal burn injuries.
* Patients will be diagnosed with median nerve conduction study and Phalen sign and tinel test.
* Patients age: 20 to 60 years

Exclusion Criteria:

* Patients with severe (absent sensory or motor waves) and mild (sensory nerve latency >3.5 ms at third digit) CTS according to EMG-NCV study.
* Conditions that could impact upon or impacted by outcome measures or laser intervention (e.g. hypothyroidism, cancer, active infection, pulmonary disease, acquired immunodeficiency syndrome, associated myopathy, myelopathy, history of neck and/or shoulder surgery, drugabuse, corticosteroids consumption, and pregnancy)
* Patients received continuous physical therapy or exercise during the previous two weeks or taking analgesic or anti-inflammatory drugs during the week prior to the baseline assessment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity. | 2 months
  Intensity of pain will be measured by visual analogue scale at baseline and at the end of the 3months. Visual analogue scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity

SECONDARY OUTCOMES:
Symptoms and Functions. | 2 months
  Boston Carpal Tunnel Questionnaire (BCTQ) The BCTQ evaluates the severity of symptoms and the functional status of patients with carpal tunnel syndrome. The symptom severity scale (SSS) consists of 11 questions covering symptom severity including night and day numbness, pins and needles, pain, and muscle weakness and scores from 1 point (mildest) to 5 points (most severe). The functional status scale (FSS) consists of 8 points concerning the patient's problems in performing specific activities such as writing, holding a book, buttoning up the shirt, holding the phone, opening jam jar, doing hard house chores, taking a bath, carrying a shopping bag, and dressing ranging from 1 point (no difficulty with the activity) to 5 points (cannot perform the activity at all). The higher the score, the greater the severity of the symptoms, and the disability of the patient would be
Median Nerve conduction Study | 2 months
  median nerve conduction study will be measured at the base line and at the end of the treatment period of two months.
Muscle strength assessment | 2 Months
  will be measured using the hand held daynamo-meter at the beginning and at the end of 2 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared after six months ofpublication.
Access Criteria: Study Protocol Study results